CLINICAL TRIAL: NCT06751303
Title: Patient Preferences for Precision Medicine
Brief Title: Patient Preferences for Precision Medicine: Determining Optimal Patient Quality of Life Using PARPi's
Acronym: 4PDQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Laura Hopkins, Professor of Oncology, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4118
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer; Quality of Life
Keywords: PARPi; HRD testing
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a pragmatic trial which offers HRD testing and for patients HRProficient, a patient decision aid to help them decide whether niraparib is right for them. Whatever they decide, we followup with QoL questionnaires and assessment of time to progression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRD Tested (Other): HRP patients are given a decision aid, while HRD patients are not given a decision.
  Interventions: Other: Patients that are HRP are given a decision aid for PARPi use

INTERVENTIONS:
Other: Patients that are HRP are given a decision aid for PARPi use — Study created patient decision aid if the first for HRD tested Ovarian Cancer patients

SUMMARY:
Patients with ovarian cancer with defective DNA repair mechanisms derive substantial benefit from PARP inhibitor (PARPi) maintenance therapy. Both niraparib and olaparib are effective inhibitors of PARP, which exploit already defective DNA repair mechanisms (e.g., via BRCA mutations), particularly those with homologous recombination deficiency (HRD). These two PARPis have notably different toxicity profiles, with niraparib showing many more severe side effects. In this Ovarian Cancer Canada funded study, we will implement perform HRD testing for ovarian cancer patients in Saskatchewan with response to platinum-based chemotherapy. This information will provide personalized and precision estimates about the amount of benefit that can be expected from taking a PARPi. We will evaluate both treatment outcomes and quality of life in a real-world study setting, to inform future decision-making regarding efficacy, quality of life and cost-effectiveness of PARPi therapy, specifically for niraparib.

We hypothesize that for patients who are homologous recombinant proficient (HRP), the median 32.7-month incremental benefit (in delaying cancer progression) from taking a PARPi (niraparib is the only PARPi approved in this setting) will not be seen as being value-add when balanced by the decreased quality of life that accompanies the first 6-12 weeks of therapy. We also hypothesize that for women who are HRP, that PARPi therapy will not be cost-efficient.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected stage 3/4 high grade serous or endometrioid ovarian cancer Able to provide oral consent and complete questionnaires in English as per study protocol

Exclusion Criteria:

* Ineligible for Maintenace PARPi therapy Refusal to undergo HRD testing

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-17 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2027-09-16 (Estimated)

PRIMARY OUTCOMES:
Patient decision for use of PARPi therapy | 6 Monhs
  The proportion of HRP patients who choose to undergo PARP therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Saskatchewan Cancer Center, Saskatoon, S, Canada

IPD SHARING:
Plan to Share IPD: No